CLINICAL TRIAL: NCT01927848
Title: Improving Gait in Persons With Knee Related Mobility Limitations by Rosenoids® Food Supplement: a Randomized Double-blind Placebo-controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Marius Henriksen, Senior Researcher, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 127
Record Dates: First submitted 2013-08-16; First posted 2013-08-23 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Knee Related Walking Limitations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosehip (Experimental): Dosage: 3 capsules once daily with meals (daily dose: 2.25 g powder).
  Interventions: Dietary Supplement: Rosehip
- Placebo (Placebo Comparator): Dosage: 3 capsules once daily with meals
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Rosehip — Rosehip powder made from the fleshy orange walls (hypanthiums) of Rosehips with the achenes (seeds) removed, from the wild growing species Dog Rose (Rosa canina L.), in addition to vitamin C as sodium ascorbate. The active ingredient complex is Rosenoids®, Vitamin C, flavonoids, carotens, triterpene acids, and galactolipids. Rosenoids® is the registered name for the bioactive complex isolated from the rose-hip (Rosa canina) used in RH01. It is being supplied as capsules containing 750 mg of the Rosehip powder and 26.7 mg vitamin C.
  Arms: Rosehip
Dietary Supplement: Placebo — The placebo used in this study will be identical to the Rosehip capsules in both appearance and taste, except that it will not contain the active Rosehip powder ingredient Rosenoids® or vitamin C.
  Arms: Placebo

SUMMARY:
Knee related mobility limitations are the leading cause of disability in the western world. It is a very expensive and debilitating condition when the cost of lost productivity and personal assistance is considered.

In recent years there has been a growing interest in alternative medicine and many individuals seek such treatments. Rosehip, that is sold as a nutritional supplement, has been particular popular, and has been shown effective in relieiving pain - albeit the evidence is scarce.

The purpose of this study is to evaluate the efficacy of specialized rosehip powder nutritional additives (Rosenoids®) on knee joint function during walking in subjects with knee-related walking limitations.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 40
* Self-reported knee-related walking disability
* In general good health, in the opinion of the Investigator, based on medical history and physical examination and, if necessary, laboratory values. Laboratory tests are prescribed by the Investigator at the screening visit.
* A body mass index (BMI) of ≤35 kg/m2
* Speaks, reads and writes Danish language

Exclusion Criteria:

* Usage of Rosehip nutritional supplements within the last 3 months
* History of symptoms of autoimmune disorders.
* Planned surgical procedure during the duration of the study
* History, diagnosis, or signs and symptoms of clinically significant neurological disease
* Alcohol or drug abuse within the last 5 years
* History, diagnosis, signs or symptoms of any clinically significant psychiatric disorder
* Subjects with regional pain syndromes suggestive of lumbar compressions with radiculopathy or at risk of developing radiculopathy.
* Any other condition, which in the opinion of the Investigator, would put the subject at increased safety risk or otherwise make the subject unsuitable for this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Knee joint biomechanics during walking | 12 weeks
  3-D kinematic gait data is obtained using a 6-camera Motion Analysis System sampling at 100 Hz capturing positions and movements of reflective markers placed on the skin and arranged in the Plug-in-Gait configuration. Ground reaction forces and moments are obtained with two 6-channel force platforms (Advanced Mechanical Technologies, Inc., Newton, MA, USA) operating at 1500 Hz synchronized with the camera system. Specialized software is used to generate lower extremity angular kinematic and kinetic data using inverse dynamics.

SECONDARY OUTCOMES:
Circulating levels of C-reactive protein (blood samples) | 12 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | week 12
  A questionnaire with suggestive leading questions, assessing adverse events at large - not necessarily adverse effects in a generic framework using options based on standards applied previously is used.
Physician global assessment of patient disease | week 12
  Physician's global assessment of overall health at clinical visits is scored on a 100 mm visual analogue scale (VAS)
Self-reported status of the participants' knee and associated problems | week 12
  Knee Osteoarthritis and Injury Outcome Score (KOOS)
Self-reported health and well-being | week 12
  Self-reported questionnaire.
Circulating levels of Alanine AminoTransferase (blood samples) | 12 weeks
Circulating levels of Alkaline Phosphatase (blood samples) | 12 weeks

OTHER OUTCOMES:
Capsule count | week 12
  Number of capsules returned in relation to number of capsules provided.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, PhD, Principal Investigator — Parker Institute, Frederiksberg Hospital
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Ginnerup-Nielsen E, Christensen R, Bliddal H, Zangger G, Hansen L, Henriksen M. Improved gait in persons with knee related mobility limitations by a rosehip food supplement: A randomized, double-blind, placebo-controlled trial. Gait Posture. 2015 Sep;42(3):340-7. doi: 10.1016/j.gaitpost.2015.07.001. Epub 2015 Jul 19. PMID 26234471